CLINICAL TRIAL: NCT06624423
Title: Effect of Corn Silk Tea on Hypertension
Acronym: CST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pir Mehr Ali Shah Arid Agriculture University (Other)
Responsible Party: Principal Investigator, Aimon Batool, Principle Investigator Aimon, Pir Mehr Ali Shah Arid Agriculture University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 6087Cornsilk
Record Dates: First submitted 2024-09-22; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): Control Group treated with only antihypertensive medications
- Treatment group 1 (Experimental): T1 group treated with 2g of Corn Silk Tea twice per day.
  Interventions: Other: corn silk tea
- Treatment group 2 (Experimental): T2 group treated with 4g of Corn Silk tea twice per day
  Interventions: Other: corn silk tea

INTERVENTIONS:
Other: corn silk tea — Corn Silk Tea
  Arms: Treatment group 1; Treatment group 2

SUMMARY:
Subjects having hypertension were divided into 3 groups. one control and two experimental who were provided with 2g and 4g of corn silk tea twice per day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Subjects with Hypertension both male and female Subjects above age 30 years

-

Exclusion Criteria:

* Subjects below age 30 years Pregnant and Lactating women Subjects with no co morbidities

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 12 weeks
  Diastolic and Systolic blood pressure will be measured using a calibrated sphygmomanometer or an automatic digital blood pressure monitor.
  Measurements will be taken in a seated position after the participant will have rested for at least 5 minutes.
  Three readings will be taken at intervals of 1-2 minutes, and the average of these readings will be recorded to ensure accuracy.

SECONDARY OUTCOMES:
Lipid Profile | 12 weeks
  Blood samples will be collected after an 8-12 hour overnight fast. Lipid profile will be measured using standard biochemical assays (such as enzymatic colorimetric methods) in a clinical laboratory. Total cholesterol, Low-Density Lipoproteins, High-Density Lipoproteins and Triglycerides were measured.
Anthropometric Measurements | 12 weeks
  Body mass measurements and waist circumference will be measured. BMI will be calculated by measuring height and weight using a standard stadiometer and weighing scale,and applying the formula. BMI=weight in kg/height in m2 Waist circumference (WC) will be measured using a non-stretchable measuring tape, placed directly on the skin at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest

CONTACTS AND LOCATIONS:
Overall Officials: Asma Sohail, Ph.D. Food Technology, Principal Investigator — Pir Mehr Ali Shah Arid Agriculture University
Locations (1):
- Institute of Food and Nutritional Sciences, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No